CLINICAL TRIAL: NCT06148519
Title: Comparing Preschool-Aged Refractive Measurements and Amblyopia Risks Using the 2WIN-S Portable Refractor with Vision Screening by Cycloplegic Refraction in Bangkok
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because the research team plans to change the protocol, we do not plan to conduct cycloplegic refraction, which requires dilation. Instead, we will use only 2-WINS for eye and vision screening. Additionally, we will change the study site
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 162/2566
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2023-11

CONDITIONS: 2WIN-S Portable Refractor
Keywords: Refraction; vision screening; preschool aged children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Using 2WIN-S portable refractor for amblyopia screening (Experimental)
  Interventions: Diagnostic Test: 2WIN-S portable refractor

INTERVENTIONS:
Diagnostic Test: 2WIN-S portable refractor — All participants will be tested by 2WIN-S portable refractor without eye dilatation. If the 2WIN-S reports non-referral, participant will be tested visual acuity by optometrist. If the 2WIN-S reports referral, participant will be tested cycloplegic refraction by pediatric ophthalmologist, then tested by 2WIN-S again. The participant whose result is abnormal will be referred to the hospital for further management.

SUMMARY:
The goal of this diagnostic test is to compare the results of refraction and amblyopia risks between using 2WIN-S portable refractor and cycloplegic refraction in pre-school age.

All participants will be tested by 2WIN-S portable refractor.

ELIGIBILITY:
Inclusion Criteria:

* corrected visual acuity 0.1 logMAR (Snellen 20/25) or better
* Age 3-6 years old who studies in the kindergarten school that joins the study
* Parents sign informed consent form about allowing their child to join the study

Exclusion Criteria:

* other eye conditions causing visual and 2WIN-S portable refractor working disturbance such as media opacity, history of ocular surgery, strabismus, etc.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Significant refractive errors defined by AAPOS | At baseline.
  Measuring spherical equivalent(SE) and cylinder(Cy), and axis to detect specific target levels of ARFs and visually significant refractive errors, as defined by AAPOS.

SECONDARY OUTCOMES:
Diagnostic accuracy for Amblyopia | At baseline.
  Diagnostic accuracy for Amblyopia, measuring by 2WIN-S device and pediatric ophthalmologist.

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No